CLINICAL TRIAL: NCT02756078
Title: Clinical Performance Evaluation of Two Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5816
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (TEST / CONTROL wear sequence) (Active Comparator): Subjects randomly assigned to the TEST Contact Lens or the CONTROL Contact Lens in the TEST / CONTROL wearing sequence will wear each of the study lenses for 4 weeks according to the manufacturer's guidelines. Subjects will be dispensed the other (second) lens type at the second dispense visit.
  Interventions: Device: TEST Contact Lens; Device: CONTROL Contact Lens
- Group 2 (CONTROL / TEST wear sequence) (Active Comparator): Subjects randomly assigned to the TEST Contact Lens or the CONTROL Contact Lens in the CONTROL / TEST wearing sequence will wear each of the study lenses for 4 weeks according to the manufacturer's guidelines. Subjects will be dispensed the other (second) lens type at the second dispense visit.
  Interventions: Device: TEST Contact Lens; Device: CONTROL Contact Lens

INTERVENTIONS:
Device: TEST Contact Lens
  Other Names: senofilcon A
Device: CONTROL Contact Lens
  Other Names: samfilcon A

SUMMARY:
This is a randomized, double-masked dispensing study where subjects will randomized into one of two lens sequences to wear each of two contact lens types for a 4-week period with each lens type.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be between 18 and 40 years of age.
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.50 Diopters (D) to -8.00 D in each eye.
* The subject's refractive cylinder must be no more than -1.00 D cylindrical correction in each eye after vertexing to the corneal plane.
* The subject must have best corrected visual acuity of 0.20 or better in each eye.
* The subject must be a current wearer of daily, spherical, soft contact lenses (no bifocal or multifocal contact lenses, no extended wear or monovision) for at least 5 days/week and at least 8 hours/day during the month prior to enrollment.
* The subject must be using digital devices (any combination of computers, tablets, smart phones etc.) for at least 8 hours over the course of a typical day.
* The subject should own a wearable pair of spectacles and wear them the day of the baseline visit.
* The subject must have normal eyes with no evidence of abnormality or disease that in the opinion of the investigator would contraindicate contact lens wear.
* The subject must meet normal eligibility conditions of binocular vision tests.
* The subject may not have any double vision at near with their habitual contact lens correction.

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear (at the investigator's discretion).
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the investigator's discretion).
* Use of any medication that causes side effects similar to side effects experienced when using digital devices, such as a subject reporting headaches associated with birth control pills (at the investigator's discretion).
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease.
* Any active ocular infection.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.).
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any known hypersensitivity or allergic reaction to the study products.
* Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 subjects were enrolled into this study. Of the enrolled, 171 subjects were randomized and dispensed at least one study lens. Of the dispensed subjects, 127 completed the study while 44 subjects were discontinued.
Groups:
- Senofilcon A/Samfilcon A: All subjects that received the senofilcon A lens during the first period and the samfilcon A lens during the second period.
- Samfilcon A/Senofilcon A: All subjects that received the samfilcon A lens during the first period and the senofilcon A lens during the second period.
Period: Period 1
Arm/Group | Senofilcon A/Samfilcon A | Samfilcon A/Senofilcon A
Started | 85 | 86
Completed | 76 | 64
Not Completed | 9 | 22
Not completed — Unsatisfactory Lens Fitting | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 10
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Lens Discomfort | 2 | 2
Period: Period 2
Arm/Group | Senofilcon A/Samfilcon A | Samfilcon A/Senofilcon A
Started | 76 | 64
Completed | 70 | 57
Not Completed | 6 | 7
Not completed — Adverse Event | 3 | 5
Not completed — Unsatisfactory Lens Fitting | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled in the study, i.e. signed informed consent form.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.9 (4.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 78
  Black or African American | 1
  White | 114
  Other | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 200

OUTCOME MEASURES:

1. Primary Outcome: Overall CLUE Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Senofilcon A: All subjects that wore the senofilcon A lens during either the first or second period of the study.
- Samfilcon A: All subjects that wore the samfilcon A lens during either the first or second period of the study.
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
Units on a Scale | 65.0 (22.47) | 60.3 (23.71)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE score; Bayesian hierarchical model; A 98% credible interval for the posterior mean difference was used to demonstrate non-inferiority between the senofilcon A and samfilcon A lenses; Posterior Mean Difference = 5.0, 98% CI 2-sided [1.30 to 8.73], Standard Deviation 1.796 — Mean difference was calculated as Test (senofilcon A) minus Control (samfilcon A)

2. Secondary Outcome: Overall CLUE Handling
Description: Overall Handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
Units on a Scale | 66.7 (18.58) | 52.9 (22.99)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE score; Bayesian hierarchical model; A 95% credible interval for the posterior mean difference was used to demonstrate non-inferiority between the senofilcon A and samfilcon A lenses; Posterior Mean Difference = 13.7, 95% CI 2-sided [10.34 to 17.05], Standard Deviation 1.701 — Mean difference was calculated as Test (senofilcon A) minus Control (samfilcon A)

3. Secondary Outcome: Time to Haze
Description: Time to haze measure the maximum time a contact lens wearers can keep their eye open without their vision becoming hazy. It was a measure of how the drying of the contact lens surface with open eyes affects vision.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
seconds | 9.4 (5.01) | 9.7 (5.65)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -2 hour was used; Bayesian hierarchical model; [statistical method as in outcome 2, analysis 1]; Posterior mean difference = -0.37, 95% CI 2-sided [-1.00 to 0.25], Standard Deviation 0.313; Mean difference was calculated as senofilcon A minus samfilcon A

4. Secondary Outcome: Average Wear Time
Description: Average lens wear time with the study lenses were recorded in hour at each follow-up visit.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
Hours | 11.5 (3.57) | 11.55 (3.57)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -2 hour was used; Bayesian hierarchical model; [statistical method as in outcome 2, analysis 1]; Posterior mean difference = -0.06, 95% CI 2-sided [-0.27 to 0.16], Standard Deviation 0.107 — Mean difference was calculated as senofilcon A minus samfilcon A

5. Secondary Outcome: Average Comfortable Wear Time
Description: Average comfortable lens wear time with the study lenses were recorded in hour at each follow-up visit.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
Hours | 9.6 (3.73) | 9.6 (3.86)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -2 hour was used; Bayesian hierarchical model; [statistical method as in outcome 2, analysis 1]; Posterior mean difference = 0.05, 95% CI 2-sided [-0.47 to 0.57], Standard Deviation 0.261 — Mean difference was calculated as senofilcon A minus samfilcon A

6. Secondary Outcome: Difference in Total Device Use Time and Comfortable Wear Time During Device Use
Description: Subjects reported the total duration of their digital device use and comfortable lens wear time during digital device use.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
Hours | 1.2 (1.74) | 1.2 (1.81)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of -2 hour was used; Bayesian hierarchical model; [statistical method as in outcome 2, analysis 1]; Posterior mean difference = -0.05, 95% CI 2-sided [-0.36 to 0.26], Standard Deviation 0.159 — Mean difference was calculated as senofilcon A minus samfilcon A

7. Secondary Outcome: Comfort at the End of the Day
Description: Subjects graded the comfort level at the end of the day using 5- point scale (1=excellence, 2=very good, 3=good, 4=fair and 5=poor). The average end of day comfort grade was reported for each lens type.
Time Frame: Up to 4-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Samfilcon A
Number analyzed (Participants) | 127 | 127
units on a scale | 2.6 (1.21) | 2.7 (1.26)
Statistical Analysis 1: Comparison: Senofilcon A vs Samfilcon A; Test type: Non-Inferiority — A non-inferiority margin of 0.67 was used; Bayesian multinomial model; A 95% credible interval for the posterior odds ratio was used to demonstrate non-inferiority between the senofilcon A and samfilcon A lenses; Posterior odds ratio = 1.35, 95% CI 2-sided [0.99 to 1.79], Standard Deviation 0.203 — Odds ratio was calculated as senofilcon A over samfilcon A

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 8 weeks per subject.
Groups:
- Samfilcon A: All subjects that wore the samfilcon A lens during either period of the study.
Arm/Group | Senofilcon A | Samfilcon A
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/171
Other Adverse Events (participants affected / at risk) | 18/171 | 29/171
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=171) | Samfilcon A (N=171)
Non-significant Infiltrative Event (Eye disorders) | 6 (10) | 2 (2)
Non-significant Allergic Conjunctivitis (Eye disorders) | 0 (0) | 3 (5)
Non-significant - Swollen Caruncle (Eye disorders) | 0 (0) | 1 (1)
Non-significant Conjunctival Redness and Staining (Eye disorders) | 0 (0) | 5 (5)
Non-significant Bulbar Redness (Eye disorders) | 0 (0) | 1 (1)
Non-significant Grade 3-4 Conjunctival Staining (Eye disorders) | 0 (0) | 2 (3)
Non-significant Symptoms, Problems or complaints requiring treatment (Eye disorders) | 0 (0) | 1 (2)
Non-significant Bacterial Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Non-significant Keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Non-significant Limbal Nodules (Eye disorders) | 0 (0) | 1 (2)
Non-significant Foreign Body (Eye disorders) | 1 (1) | 0 (0)
Stye (Eye disorders) | 1 (1) | 0 (0)
Non-significant Bulbar and Limbal Redness (Eye disorders) | 0 (0) | 4 (5)
Non-significant Localized Allergic Reaction (Eye disorders) | 2 (5) | 0 (0)
Non-significant Corneal Tissue Overgrowth (Eye disorders) | 1 (1) | 0 (0)
Non-significant slit lamp finding Grade 2 or less requiring treatment (Eye disorders) | 0 (0) | 1 (1)
Non-significant Conjunctival Redness Grade 3 or Higher (Eye disorders) | 0 (0) | 1 (2)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Non-significant Reaction to Eye Drop (Eye disorders) | 0 (0) | 1 (2)
Flu (Immune system disorders) | 1 (1) | 1 (1)
Non-significant Phlyctenules (Eye disorders) | 0 (0) | 1 (1)
Stomach Flu (Immune system disorders) | 0 (0) | 1 (1)
Non-significant Superficial Deposits (Eye disorders) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Non-significant Blurred Central Vision (Eye disorders) | 0 (0) | 1 (1)
Non-significant Superior Arcuate (Eye disorders) | 1 (1) | 0 (0)
Non-significant Localized Corneal Staining (Eye disorders) | 1 (1) | 0 (0)
Non-significant Ocular Discomfort (Eye disorders) | 1 (1) | 1 (2)
Non-significant Redness (Eye disorders) | 0 (0) | 1 (1) — Patient Reported.
Non-significant Difficulty opening eye (Eye disorders) | 1 (1) | 0 (0)
Non-significant Stye (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT02756078/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02756078/SAP_001.pdf